CLINICAL TRIAL: NCT06618300
Title: Streamlined Resin Y90 Radiation Segmentectomy for Small HCC: One&Done Trial
Brief Title: Streamlined Resin Y90 Radiation Segmentectomy for Small HCC
Acronym: One&Done
Status: Enrolling by invitation | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Sirtex, Wodburn, MA (Unknown)
Responsible Party: Sponsor
Other Study IDs: LCCC2401
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: radioembolization; Yttrium-90; workflow
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Yttrium-90 (Y90) radioembolization: Patients with small Hepatocellular Carcinoma undergoing Yttrium-90 (Y90) radioembolization.

SUMMARY:
This single-arm feasibility study evaluating the safety and efficacy of streamlining Yttrium-90 (Y90) radioembolization workflow for patients with small Hepatocellular Carcinoma (<5cm) that have no aggressive features on baseline imaging. This study aims to recruit N=30 patients prospectively and consolidate the current workflow of 2 days of procedures (1st-day mapping angiography followed by nuclear medicine hepatic lung shunt fraction (LSF) calculation using Tc99-MAA planar and SPECT/CT, and 2nd-day Y90 radioembolization followed by nuclear medicine Y90 SPECT/CT) into 1-day procedure. Several studies have shown that hepatic LSF for HCC tumors smaller than 5cm in the absence of macrovascular invasion and portosystemic shunt placement is invariably <10%. Therefore, the LSF calculation can be safely omitted from the complex workflow of these patients. This study aims to illustrate that this can be done safely and efficaciously to reduce unnecessary patient travel and healthcare resource utilization. Overall, a total of 30 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has focal Hepatocellular Carcinoma and is deemed to benefit from Yttrium-90 radioembolization by the institutional multidisciplinary tumor board

Exclusion Criteria:

* All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.
* The presence of trans-jugular intrahepatic portosystemic shunt
* Total bilirubin level > 3.0 mg/dL
* Serum albumin level < 2.5 g/dL
* Aspartate and alanine aminotransferase levels no greater than five times the normal level
* Life expectancy < 12 weeks
* Eastern Cooperative Oncology Group performance status > 2
* Patients with chronic lung disease requiring supplemental oxygen at baseline or baseline SpO2 of <92%
* Patients that have tumors with central anatomical locations close the hepatic hilum or caudate lobe.
* Patients with macrovascular invasion on baseline imaging
* Known hypersensitivity to iodinated contrast agents or to any component of iodinated contrast agents refractory to standard medications (antihistamines, steroids)
* Impaired kidney function (glomerular filtration rate < 30 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine β-HCG results, obtained within 48 hours prior to the treatment or on the basis of patient history, e.g.: tubal ligation, hysterectomy or a minimum of 1 year without menses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with small Hepatocellular Carcinoma receive Yttrium-90 (Y90) radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The treatment timeline | 3 days
  The treatment timeline will be measured in days from the date of the initial consultation of the patient in the interventional radiology clinic to the date of the Yttrium-90 (Y90) radioembolization procedure.
Cumulative charges and reimbursement | 3 days
  To observe cumulative charges and reimbursement for streamlined Yttrium-90 (Y90) radioembolization treatment, billing, and reimbursement information will be obtained through the billing department. The costs will be reported in US dollars.

SECONDARY OUTCOMES:
Duration of response | 12 months
  Duration of response in the treated area and elsewhere in the liver will be recorded. The response will be categorized as objective response vs no response based on mRECIST criteria and the percentage of patients achieving clinical success will be recorded.
The safety of streamlined Y90 radioembolization | 1, 3, 6, and 12 months post Y90 radioembolization
  To demonstrate the safety of streamlined Y90 radioembolization segmental treatment for small Hepatocellular Carcinoma (HCC) by observing the incidence of radiation-induced pneumonitis and liver toxicity. Clinical and biochemical toxicity will be well documented using Common Terminology for Adverse Events Version 5, 6,7 a
Response to streamlined Y90 | 12 months
  To evaluate the efficacy of streamlined Y90 TARE for small Hepatocellular Carcinoma (HCC) using modified Response Evaluation for Solid Tumors (m-RECIST) and duration of response in the treated area and elsewhere in the liver at 12 months post-Y90. Efficacy will be categorized as objective response vs no response based on mRECIST criteria and the percentage of patients achieving clinical success will be recorded.
Hepatic lung shunt fraction | 3 days
  Hepatic lung shunt fraction (LSF) will be calculated using post-Yttrium-90 (Y90) radioembolization single photon emission computed tomography (SPECT) fused with computed tomography (CT) (SPECT/CT).

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Yu, MD, FSIR, Principal Investigator — UNC Department of Radiology
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials